CLINICAL TRIAL: NCT03992079
Title: A Single Institutional Randomized Controlled Trial for A Multimodal Enhanced Recovery Program in Anorectal Surgery
Brief Title: A Multimodal Enhanced Recovery Program in Anorectal Surgery
Acronym: ARSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is no longer at institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAS3302
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Disorders; Anorectal Disorder; Patient Satisfaction; Pain, Postoperative; Opioid Use; Opioid Abuse; Opioid Dependence
MeSH Terms: conditions — Rectal Diseases; Patient Satisfaction; Pain, Postoperative; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: After providing written informed consent, patients will be randomly assigned in a 1:1 ratio to either the control group, which uses physician preference for pain control, and generally relies on extended opioids or the experimental group, which includes preemptive pain control, targeted education, and multimodal opioid-sparing pain management during the intraoperative and postoperative periods.
Who Masked: Care Provider, Investigator
Masking Description: Randomization will be conducted by means of a secure website (Sealed Envelope), with block randomization to help balance the groups by the procedures performed within each arm. The patients, post-anesthesia care unit (PACU) staff, and study investigators performing follow up assessments, collecting, and analyzing the data will be unaware of the treatment assignments. It is not feasible to blind the operating team or site enrolment personnel as different preoperative and discharge information, medication and patient education will be given to the experimental and control groups. A numbered, sealed envelope, corresponding to the patient's assigned study number, will be opened, and the research coordinator will alert the surgeon to the patient's group assignment. Using the assumption that patients do not know the difference between enhanced recovery and usual care, the patient will not be informed of which arm they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive standard preoperative and postoperative directions, with the anesthesiologist and surgeon's preferences for analgesia during and after surgery.
- Experimental (Experimental): The experimental group will receive routine directions for surgery and a ReCOVER patient education document on the Enhanced Recovery protocol, with instructions on preoperative preparation, postoperative wound care, pain management, preventing and managing constipation, activity limitations, and return precautions. The information sheet will be provided to patients in clinic and reviewed with a member of the healthcare team to ensure an understanding of the plan.
  Interventions: Procedure: ReCOVER Enhanced Recovery Protocol

INTERVENTIONS:
Procedure: ReCOVER Enhanced Recovery Protocol — The experimental group will receive preemptive pain management before surgery, an opioid-free strategy during surgery, and an opioid-sparing multimodal pain management protocol after surgery.
  Arms: Experimental

SUMMARY:
The goal of this study is to establish whether an opioid-sparing Enhanced Recovery After Surgery (ERAS) program in ambulatory anorectal surgery can be safely introduced at a single tertiary referral center without an increase in postoperative pain or negative impact on the patient experience. A single-center, single-blinded randomized control trial is proposed, where patients will be assigned in a 1:1 ratio to either usual care, which includes extended opioids (control group) or the enhanced recovery group (experimental), which includes preemptive pain control, targeted education, and multimodal opioid-sparing pain management during the intraoperative and postoperative periods. The expected outcome is that the enhanced recovery program will significantly reduce opioid utilization with comparable pain scores and patient satisfaction after anorectal surgery.

DETAILED DESCRIPTION:
There is an opioid epidemic in the United States, and the epidemic continues to worsen. The rate of opioids prescribed, distributed, and deaths from opioid overdoses continue to increase steadily. Opioids also have the costs of abuse, dependence, diversion of unused medication, and can serve as a gateway to other illegal substances. Opioid use often begins with treatment of acute postoperative pain, and the surgical episode can be a 'gateway' to the opioid crisis. Opioids remain ubiquitous in patients undergoing surgical procedures. Among opioid-naïve patients, persistent use after surgery occurs in 6-10%.

Ambulatory surgery cases are rarely mentioned in the context of this public health crisis, but are a major contributor to the problem. Opioids are ubiquitous after ambulatory anorectal surgery and prescribed in large quantities, often several times more than what is needed or taken by patients. As patients take a fraction of the opioids prescribed, this adds to issues of opioid diversion. In colorectal surgery, ambulatory anorectal procedures are common and frequent procedures, with the potential to impact a large number of patients when implementing quality improvement. Thus, study into ERAS and ways to reduce opioids after ambulatory anorectal surgery is warranted.

This application challenges the notion that inpatient surgery should be the only target for enhanced recovery and opioid interventions. It seeks to shift the clinical practice paradigm that extended opioids are necessary after ambulatory anorectal surgery. This new application of ERAS to ambulatory anorectal surgery could address a critical barrier to progress in reducing opioids in procedures that are common but underrepresented in current research.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom surgery is planned via an anorectal approach for hemorrhoids, fissures, or fistula disease.

Exclusion Criteria:

* Patients are not eligible if currently or chronically (more than 7 days prior to presentation) on opioid medication or opioid-receptor antagonist medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Rate of Opioid Use | Up to 30 days post surgery
  Postoperative opioid use will be measured in morphine milligram equivalents per day (MME)

SECONDARY OUTCOMES:
Pain Score on the Visual Analog Scale (VAS) | Up to 30 days post surgery
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain (score of 0) and the other end meaning the worst pain imaginable (score of 100). Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Pain Score on the Functional Pain Scale (FPS) | Up to 30 days post surgery
  The Functional Pain Scale (FPS) was developed in 2001 to evaluate the effect of pain on patient function for various different types of pain. The scale ranges from 0-5 and the participants score will fall within this range 0-5 range based a combination of their subjective rating of pain and their objective opinion about how that pain interferes with daily activities. A lower score is linked to lower levels of pain and reduced interference from pain on daily activities.
Score on the EQ-5D-3L | Up to 30 days post surgery
  The EQ-5D-3L queries across five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has levels ranging from no problems (score of 1) to extreme problems (score of 5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The final "score" is coded based on the 5 responses.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah S. Keller, MS, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Tan M, Law LS, Gan TJ. Optimizing pain management to facilitate Enhanced Recovery After Surgery pathways. Can J Anaesth. 2015 Feb;62(2):203-18. doi: 10.1007/s12630-014-0275-x. Epub 2014 Dec 10. PMID 25501696
- [Background] Carmichael JC, Keller DS, Baldini G, Bordeianou L, Weiss E, Lee L, Boutros M, McClane J, Feldman LS, Steele SR. Clinical Practice Guidelines for Enhanced Recovery After Colon and Rectal Surgery From the American Society of Colon and Rectal Surgeons and Society of American Gastrointestinal and Endoscopic Surgeons. Dis Colon Rectum. 2017 Aug;60(8):761-784. doi: 10.1097/DCR.0000000000000883. No abstract available. PMID 28682962
- [Background] Swarup A, Mathis KA, Hill MV, Ivatury SJ. Patterns of opioid use and prescribing for outpatient anorectal operations. J Surg Res. 2018 Sep;229:283-287. doi: 10.1016/j.jss.2018.04.005. Epub 2018 May 9. PMID 29937003
- [Background] Rose KR, Christie BM, Block LM, Rao VK, Michelotti BF. Opioid Prescribing and Consumption Patterns following Outpatient Plastic Surgery Procedures. Plast Reconstr Surg. 2019 Mar;143(3):929-938. doi: 10.1097/PRS.0000000000005351. PMID 30817667
- [Background] Harris K, Curtis J, Larsen B, Calder S, Duffy K, Bowen G, Hadley M, Tristani-Firouzi P. Opioid pain medication use after dermatologic surgery: a prospective observational study of 212 dermatologic surgery patients. JAMA Dermatol. 2013 Mar;149(3):317-21. doi: 10.1001/jamadermatol.2013.1871. PMID 23682368
- [Background] Bates C, Laciak R, Southwick A, Bishoff J. Overprescription of postoperative narcotics: a look at postoperative pain medication delivery, consumption and disposal in urological practice. J Urol. 2011 Feb;185(2):551-5. doi: 10.1016/j.juro.2010.09.088. Epub 2010 Dec 18. PMID 21168869
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Kenan K, Mack K, Paulozzi L. Trends in prescriptions for oxycodone and other commonly used opioids in the United States, 2000-2010. Open Med. 2012 Apr 10;6(2):e41-7. Print 2012. PMID 23696768
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers---United States, 1999--2008. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1487-92. PMID 22048730
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Florence CS, Zhou C, Luo F, Xu L. The Economic Burden of Prescription Opioid Overdose, Abuse, and Dependence in the United States, 2013. Med Care. 2016 Oct;54(10):901-6. doi: 10.1097/MLR.0000000000000625. PMID 27623005
- [Background] Baker DW. History of The Joint Commission's Pain Standards: Lessons for Today's Prescription Opioid Epidemic. JAMA. 2017 Mar 21;317(11):1117-1118. doi: 10.1001/jama.2017.0935. No abstract available. PMID 28241189
- [Background] Kessler ER, Shah M, Gruschkus SK, Raju A. Cost and quality implications of opioid-based postsurgical pain control using administrative claims data from a large health system: opioid-related adverse events and their impact on clinical and economic outcomes. Pharmacotherapy. 2013 Apr;33(4):383-91. doi: 10.1002/phar.1223. PMID 23553809
- [Background] Lee JS, Hu HM, Edelman AL, Brummett CM, Englesbe MJ, Waljee JF, Smerage JB, Griggs JJ, Nathan H, Jeruss JS, Dossett LA. New Persistent Opioid Use Among Patients With Cancer After Curative-Intent Surgery. J Clin Oncol. 2017 Dec 20;35(36):4042-4049. doi: 10.1200/JCO.2017.74.1363. Epub 2017 Oct 19. PMID 29048972
- [Background] Carroll I, Barelka P, Wang CK, Wang BM, Gillespie MJ, McCue R, Younger JW, Trafton J, Humphreys K, Goodman SB, Dirbas F, Whyte RI, Donington JS, Cannon WB, Mackey SC. A pilot cohort study of the determinants of longitudinal opioid use after surgery. Anesth Analg. 2012 Sep;115(3):694-702. doi: 10.1213/ANE.0b013e31825c049f. Epub 2012 Jun 22. PMID 22729963
- [Background] Van Backer JT, Jordan MR, Leahy DT, Moore JS, Callas P, Dominick T, Cataldo PA. Preemptive Analgesia Decreases Pain Following Anorectal Surgery: A Prospective, Randomized, Double-Blinded, Placebo-Controlled Trial. Dis Colon Rectum. 2018 Jul;61(7):824-829. doi: 10.1097/DCR.0000000000001069. PMID 29771804
- [Background] Parrish AB, O'Neill SM, Crain SR, Russell TA, Sonthalia DK, Nguyen VT, Aboulian A. An Enhanced Recovery After Surgery (ERAS) Protocol for Ambulatory Anorectal Surgery Reduced Postoperative Pain and Unplanned Returns to Care After Discharge. World J Surg. 2018 Jul;42(7):1929-1938. doi: 10.1007/s00268-017-4414-8. PMID 29318355
- [Background] Gloth FM 3rd, Scheve AA, Stober CV, Chow S, Prosser J. The Functional Pain Scale: reliability, validity, and responsiveness in an elderly population. J Am Med Dir Assoc. 2001 May-Jun;2(3):110-4. PMID 12812581
- See also: Centers for Disease Control and Prevention. Wide-ranging online data for epidemiologic research (WONDER). Atlanta, GA: CDC, National Center for Health Statistics; 2017. — https://wonder.cdc.gov/
- See also: Center for Behavioral Health Statistics and Quality. (2017). 2016 National Survey on Drug Use and Health: Detailed Tables. Substance Abuse and Mental Health Services Administration, Rockville, MD. — https://www.samhsa.gov/data/sites/default/files/NSDUH-DetTabs-2016/NSDUH-DetTabs-2016.pdf